CLINICAL TRIAL: NCT06158568
Title: Effects of Percutaneous Electrical Nerve Stimulation and Exercise for Patients With Subacromial Pain Syndrome
Brief Title: Percutaneous Electrical Nerve Stimulation and Exercise for Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: César Fernández-de-las-Peñas (Other)
Responsible Party: Sponsor-Investigator, César Fernández-de-las-Peñas, Clinical Professor, Universidad Rey Juan Carlos
Organization: Universidad Rey Juan Carlos (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: URJC0609202218622
Record Dates: First submitted 2023-11-27; First posted 2023-12-06 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Shoulder Pain
Keywords: Neuromodulation; Percutaneous Nerve Stimulation; Exercise
MeSH Terms: conditions — Shoulder Pain; Motor Activity | interventions — Transcutaneous Electric Nerve Stimulation; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Percutaneous Electrical Nerve Stimulation (Experimental): Participants assigned to this group will received four sessions (once per week) of ultrasound guided percutaneous electrical nerve stimulation targeting the axillar and suprascapular nerves for 30 minutes. We will apply a biphasic compensated electrical current at a frequency of 2 Hz, a pulse width of 250 μs and intensity allowed over a pain-free motor threshold (muscle contraction). In addition, they will receive a program of exercises for the shoulder musculature for 3 weeks.
  Interventions: Other: Percutaneous Electrical Nerve Stimulation; Other: Exercise
- Placebo Percutaneous Nerve Stimulation (Placebo Comparator): Participants assigned to this group will received four sessions (once per week) of placebo ultrasound guided percutaneous electrical nerve stimulation targeting the axillar and suprascapular nerve. The electrical current will be off and no electrical current will be provided to the patient. In addition, they will receive the same program of exercises for the shoulder than the experimental group for three weeks.
  Interventions: Other: Placebo Percutaneous Electrical Nerve Stimulation; Other: Exercise
- Exercise (Active Comparator): Participants assigned to this group will receive the same program of exercises for the shoulder than the remaining groups for three weeks.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Percutaneous Electrical Nerve Stimulation — Application of a electrical current percutaneously (at the motor response intensity) targeting the suprascapular and axillar nerves
  Arms: Percutaneous Electrical Nerve Stimulation
Other: Placebo Percutaneous Electrical Nerve Stimulation — Application of sham electrical current (no intensity) percutaneously targeting the suprascapular and axillar nerves
  Arms: Placebo Percutaneous Nerve Stimulation
Other: Exercise — Application of three weeks of progressive exercises targeting the shoulder musculature

SUMMARY:
Based on the available literature, application of percutaneous electrical nerve stimulation interventions targeting peripheral nerves (also called percutaneous neuromodulation) has shown positive effects for improving pain-related and functional outcomes in musculoskeletal chronic pain. Studies investigating the use of this intervention for the shoulder are lacking.

DETAILED DESCRIPTION:
Based on the available literature, application of percutaneous electrical nerve stimulation interventions targeting peripheral nerves (also called percutaneous neuromodulation) has shown positive effects for improving pain-related and functional outcomes in musculoskeletal chronic pain. Studies investigating the use of this intervention for the shoulder are lacking.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral non-traumatic shoulder pain (positive painful arc during shoulder abduction and a positive Hawkins test on clinical examination)
* Shoulder pain from at least 3 months
* Shoulder pain of more than 3/10 points on a NPRS

Exclusion Criteria:

* Bilateral shoulder symptoms
* Younger than 18 or older than 65 years
* History of shoulder traumatisms, fractures or dislocation
* Diagnosis of cervical radiculopathy or myelopathy
* Previous interventions with steroid injections in the shoulder area
* Comorbid medical conditions, e.g., fibromyalgia syndrome
* Previous history of shoulder or neck surgery
* Any type of intervention for the neck-shoulder area during the previous year
* Fear to needles

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-04-27 (Actual)

PRIMARY OUTCOMES:
Changes in disability between baseline and follow-up periods | Baseline, one week after the last intervention and 1 and 3 months after the intervention
  The Disabilities of the Arm, Shoulder and Hand (DASH) will be used to determine the disability induced by shoulder pain

SECONDARY OUTCOMES:
Changes in shoulder pain between baseline and follow-up periods | Baseline, one week after the last intervention and 1 and 3 months after the intervention
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' mean level of shoulder pain experienced in the preceding week in the shoulder area.
Changes in sleep quality between baseline and follow-up periods | Baseline, one week after the last intervention and 1 and 3 months after the intervention
  The Pittsburgh Sleep Quality Index (PSQI) will be used to evaluate the quality of sleep
Changes in anxiety/depressive symptoms between baseline and follow-up periods | Baseline, one week after the last intervention and 1 and 3 months after the intervention
  The Hospital Anxiety and Depression Scale (HADS, A: Anxiety; D: Depression) will be used to evaluate the presence of anxiety/depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: César Fernández-de-las-Peñas, PhD, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- César Fernández-de-las-Peñas, Madrid, Rest of the World, Spain